CLINICAL TRIAL: NCT06101719
Title: Use of a Water Soluble Contrast-Based Protocol to Assist in the Management of Pediatric Adhesive Small Bowel Obstruction
Acronym: SBO
Status: Completed | Type: Observational
Sponsor: Children's Hospital Colorado (Other)
Collaborators: Children's Hospital Los Angeles (Other); University of California, San Francisco (Other); Oregon Health and Science University (Other); Rady Children's Hospital, San Diego (Other); Phoenix Children's Hospital (Other); Primary Children's Hospital (Other); Children's Medical Center Dallas (Other); Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Shannon Acker, Associate Professor, Pediatric Surgery, Children's Hospital Colorado
Other Study IDs: 20-2538
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Small Bowel Obstruction; Contrast Media Adverse Reaction
Keywords: Pediatric adhesive small bowel obstruction; enteral contrast challenge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Contrast Group: Inclusion criteria: children 1-20 years diagnosed with an adhesive small bowel obstruction by an attending pediatric surgeon and underwent a trial of nonoperative management (NOM) on hospital admission and received an enteral contrast challenge. Exclusion criteria included peritonitis, suspicion of incarcerated or internal hernia, active intra-abdominal malignancy, inflammatory bowel disease, <4 weeks since the most recent abdominal operation,45 pneumatosis, pneumoperitoneum, or known contrast allergy. If the attending surgeon made the decision to take a child directly to the operating room (OR) with no attempt at NOM, these children were excluded. Children under one year of age were excluded as the rate of successful NOM is lower in this age group
  Interventions: Diagnostic Test: Enteral contrast challenge
- No Contrast group: Inclusion criteria: children 1-20 years diagnosed with an adhesive small bowel obstruction by an attending pediatric surgeon and underwent a trial of nonoperative management (NOM) on hospital admission and who did not receive an enteral contrast challenge. Exclusion criteria included peritonitis, suspicion of incarcerated or internal hernia, active intra-abdominal malignancy, inflammatory bowel disease, <4 weeks since the most recent abdominal operation, pneumatosis, pneumoperitoneum, or known contrast allergy. If the attending surgeon made the decision to take a child directly to the operating room (OR) with no attempt at NOM, these children were excluded. Children under one year of age were excluded as the rate of successful NOM is lower in this age group

INTERVENTIONS:
Diagnostic Test: Enteral contrast challenge — Contrast agent, volume of contrast, and contrast dilution were not standardized across sites due to the differences in hospital specific formularies; otherwise, the protocol was standardized across sites. Diatrizoate meglumine (osmolality of 1940 mOsm/kg) was used preferentially at eight sites and Ioversol (702 mOms/kg) at one site. Patients received 30-200ml (based on age or weight depending on site) of enteral contrast followed by X-rays at 8-12 hours and 24 hours after contrast administration.
  Groups: Contrast Group

SUMMARY:
The goal of this prospective observational study is to evaluate the diagnostic and therapeutic utility of an enteral contrast challenge for pediatric patients with adhesive small bowel obstruction (ASBO). The aims are to

1. Determine if an enteral contrast challenge is safe in the evaluation of children with ASBO
2. Determine if an enteral contrast challenge decreases the need for operation among children with ASBO Children with ASBO who are cared for at one of 9 participating sites who undergo a trial of non operative management will be observed. Comparisons will be made between those who receive and enteral contrast challenge and those who do not. Outcomes to be evaluated include adverse events related to the contrast, rate of operative intervention, and hospital length of stay.

DETAILED DESCRIPTION:
Study Design and Patient Population The investigators conducted a prospective observational study at nine children's hospitals that are members of the Western Pediatric Surgery Research Consortium. IRB approval was obtained from each site with waiver of consent for enrollment. Enrollment took place between 2020-2022. Inclusion criteria were children 1-20 years diagnosed with an ASBO by an attending pediatric surgeon and underwent a trial of nonoperative management (NOM) on hospital admission. The use of an enteral contrast protocol was at the discretion of the attending surgeon. Exclusion criteria included peritonitis, suspicion of incarcerated or internal hernia, active intra-abdominal malignancy, inflammatory bowel disease, <4 weeks since the most recent abdominal operation, pneumatosis, pneumoperitoneum, or known contrast allergy. If the attending surgeon made the decision to take a child directly to the operating room (OR) with no attempt at NOM, these children were excluded. Children under one year of age were excluded as the rate of successful NOM is lower in this age group.

Site details and Contrast Protocols At the start of the study, four of the nine sites had a contrast protocol in place for ASBO diagnosis and management. During the course of the study, contrast protocols were developed and implemented at each of the five additional sites. At study initiation, three sites used contrast routinely, one used it selectively and 5 did not use contrast. At study conclusion, five sites used contrast routinely and four used it selectively.

Contrast agent, volume of contrast, and contrast dilution were not standardized across sites due to the differences in hospital specific formularies; otherwise, the protocol was standardized across sites. Diatrizoate meglumine (osmolality of 1940 mOsm/kg) was used preferentially at eight sites and Ioversol (702 mOms/kg) at one site. Patients received 30-200ml (based on age or weight depending on site) of enteral contrast followed by X-rays at 8-12 hours and 24 hours after contrast administration. Patients were included in the contrast arm if enteral contrast, administered as part of an abdominal CT scan, was followed with subsequent x-rays to assess for progression of contrast to the colon. Failure (complete bowel obstruction) was defined as failure of contrast having not reached the colon by 24 hours after oral administration at which point operative intervention was recommended. The decision to operate was at the discretion of the attending surgeon.

Sample Size Calculation The study was powered to detect a 15% difference in operative rate between the contrast and no contrast groups based on the adult literature. To detect this difference with 80% power, the investigators aimed to enroll 314 patients.

Data Collection and Outcomes Study data were collected and managed using the Research Electronic Data Capture (REDCap) software tool hosted at the University of Colorado. REDCap is a secure, web-based application designed to support data capture for research studies. The surgical inpatient census was monitored daily by study personnel at each site for patients with ASBO. Once identified, data were collected based on a review of the electronic medical record at each site 30 days following hospital discharge. Data collected included patient demographics, medical and surgical history, clinical presentation, laboratory studies, and imaging, management approach including type, volume, dilution of any contrast agent used. Complications specific to the contrast administration including allergic reaction, aspiration of contrast, cardiac arrhythmia, and renal failure were recorded. Details of the hospital course including length of stay, need for operation, indications for operation, and subsequent postoperative course and complications were also included.

Statistical Analysis Descriptive statistics were summarized for continuous variables with medians and interquartile ranges, and for categorical variables with frequencies and percentages. Group differences were tested via t-test or Kruskal-Wallis test for continuous variables and Chi-Squared test or Fisher's Exact test for categorical variables. Comparisons were made between those who received contrast and those who did not. Logistic regression was used to assess the association between contrast and need for operation adjusting for age, body mass index for age z-score (or weight for height z-score for patients under 24 months of age per Centers for Disease Control and Prevention standards), volume of contrast administered, and number of previous laparotomies (< 3 v. ≥3). A subset analysis was performed among patients who received enteral contrast. Comparisons were made based on type of contrast agent used and final osmolality of contrast administered. Additional comparisons were made between only those patients who were successfully managed nonoperatively and then between those patients who required abdominal operation, based on contrast status.

ELIGIBILITY:
Inclusion Criteria:

1. children 1-20 years
2. diagnosed with an adhesive small bowel obstruction by an attending pediatric surgeon
3. underwent a trial of nonoperative management on hospital admission

Exclusion Criteria:

1. peritonitis
2. suspicion of incarcerated or internal hernia
3. active intra-abdominal malignancy
4. inflammatory bowel disease
5. less than four weeks since most recent abdominal operations
6. pneumatosis
7. pneumoperitoneum
8. known contrast allergy

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with adhesive small bowel obstruction admitted to one of 9 participating sites and underwent a trial of non operative management
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who required an operation | 1 year
  operative lysis of adhesions performed due to failure of non operative management

SECONDARY OUTCOMES:
Total hospital length of stay in days | 1 year
  total hospital length of stay among patients successfully managed non operatively
Adverse events resulting from contrast administration | 1 year
  adverse events related to contrast administration

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Acker, MD, Principal Investigator — Children's Hospital Colorado
Locations (9):
- United States (9):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, Oakland, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Medical Center of Dallas, Dallas, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided